CLINICAL TRIAL: NCT04787848
Title: Role of Endogenous Opioid Peptides in HIV-associated Chronic Widespread Pain
Brief Title: Chronic Widespread Pain in HIV: Novel Mechanisms and Therapeutics
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Responsible Party: Principal Investigator, Dr. Saurabh Aggarwal, Associate Professor in the Department of Cellular and Molecular Biology, Florida International University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 300007004
Record Dates: First submitted 2021-02-25; First posted 2021-03-09 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Chronic Widespread Pain
MeSH Terms: conditions — Chronic Pain | interventions — methylnaltrexone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- HIV negative without chronic widespread pain (Experimental): 50 Participants will be randomly administered saline or RELISTOR (Individuals weighing 38-<62 kg will receive an 8 mg dose; those weighing 62-114 kg will receive a 12 mg dose; Participants weighing more than 114 kg will receive 0.15 mg/kg) in counterbalance between visit 1 and visit 2.
  Interventions: Drug: Relistor Injectable Product
- HIV negative with chronic widespread pain (Experimental): 50 Participants will be randomly administered saline or RELISTOR (Individuals weighing 38-<62 kg will receive an 8 mg dose; those weighing 62-114 kg will receive a 12 mg dose; Participants weighing more than 114 kg will receive 0.15 mg/kg) in counterbalance between visit 1 and visit 2.
  Interventions: Drug: Relistor Injectable Product
- HIV positive without chronic widespread pain (Experimental): 50 Participants will be randomly administered saline or RELISTOR (Individuals weighing 38-<62 kg will receive an 8 mg dose; those weighing 62-114 kg will receive a 12 mg dose; Participants weighing more than 114 kg will receive 0.15 mg/kg) in counterbalance between visit 1 and visit 2.
  Interventions: Drug: Relistor Injectable Product
- HIV positive with chronic widespread pain (Experimental): 50 Participants will be randomly administered saline or RELISTOR (Individuals weighing 38-<62 kg will receive an 8 mg dose; those weighing 62-114 kg will receive a 12 mg dose; Participants weighing more than 114 kg will receive 0.15 mg/kg) in counterbalance between visit 1 and visit 2.
  Interventions: Drug: Relistor Injectable Product

INTERVENTIONS:
Drug: Relistor Injectable Product — Relistor is a peripherally acting opioid receptor antagonist approved by the FDA for relief of opioid-induced constipation
  Other Names: Methylnaltrexone Bromide

SUMMARY:
To determine if decreased production or release of endogenous opioid peptides by peripheral immune cells contributes to hypersensitivity in people with HIV

DETAILED DESCRIPTION:
The prevalence of chronic widespread pain (CWP) in individuals infected with the human immunodeficiency virus (HIV-1) includes regional and widespread musculoskeletal pain of neuropathic and inflammatory nature. HIV-related CWP leads to 10x greater odds of functional impairment. However, the specific mechanisms that contribute to CWP in HIV are not understood. Thus, pharmacological and non-pharmacological approaches to mitigate CWP have had minimal benefits, contributing to an overreliance on opioids and alarming rise in addiction and overdose. The overall objective of this study is to address the gap in the knowledge of the pathogenesis of HIV-related CWP. Specifically, the role of impaired endogenous opioid synthesis/release from leukocytes in people with HIV (PWH) who self-report CWP will be explored. Leukocytes (neutrophils, monocytes/macrophages, and lymphocytes) are a rich source of opioid peptides (Met-enkephalin, dynorphin A, β-endorphin) that inhibit nociception by binding to peripheral opioid receptors. Therefore, to establish whether decreased peripheral opioid peptides correlate with experimental pain measures in PWH with self-reported CWP, quantitative sensory testing (QST) will be completed before and after administration of methylnaltrexone bromide (RELISTOR), a clinically available, peripherally acting opioid receptor antagonist.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed HIV diagnosis and currently a patient in the UAB 1917 HIV Clinic
* Age 19 - 65; the lower end of this age range was chosen to capture young adults with HIV infection, and participants over 65 years are increasingly likely to meet one or more exclusion criteria
* All people living with HIV must be currently receiving stable antiretroviral therapy (ART) for inclusion in this study
* Non-HIV participants must be confirmed as HIV negative. HIV-negative participants with chronic widespread pain must self-report bodily pain more than once per week for at least three consecutive months and HIV-negative participants without chronic pain must self-report no pain, or pain less frequently than once per week for at least three consecutive months

Exclusion Criteria:

* Anemia
* Current or past history of blood disorders which may increase hemolysis
* Active microbial infections which may alter the quantity or quality of blood inflammatory cells such as monocytes and neutrophils
* Use of certain medication other than antiretroviral therapy that might conflict with study observations. However, participants will not be excluded or asked to withdraw from medications used for pain management since temporary withdrawal from these medications could affect pain measures (exceptions will be therapies such as methadone or buprenorphine used to treat opioid addiction). Only those who are stable on these medications for at least 60 days will be included. All patient medications used for at least the 60 days prior to participation will be recorded and controlled in statistical analyses as needed
* Systemic rheumatic disease (e.g., rheumatoid arthritis, systemic lupus erythematosus). These rheumatologic conditions will be excluded due to their autoimmune characteristic. . Cachexia (wasting syndrome) and severe frailty. This exclusion is in place to protect against the stress of experimental pain testing
* A history of clinically significant surgery in the past year
* Uncontrolled hypertension (i.e. SBP/DBP of >150/95) or cardiovascular or peripheral arterial disease. These exclusions are in place primarily for safety reasons because the cold pressor task represents a cardiovascular challenge. However, uncontrolled hypertension can also affect pain perception, which is another reason for excluding these individuals
* Poorly controlled diabetes (HbA1c > 8%) for both safety reasons, and because diabetic neuropathy could alter pain perception
* Neurological disease (e.g. Parkinson's, multiple sclerosis, epilepsy)
* Serious psychiatric disorder requiring hospitalization within the past 12 months or characterized by active suicidal ideation
* Any participant deemed to be actively suicidal upon study screening will be escorted to the UAB emergency room and evaluated by the Psychiatry Service
* Diminished cognitive function that would interfere with understanding of study procedures. The Realm Health Literacy Test will be administered to ensure that participants are free of cognitive impairment that would compromise study participation
* Pregnancy. Inclusion/exclusion criteria will be verified using the screening tool in combination with review of participants' medical records

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-11-15 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Quantitative sensory testing (QST) | At baseline (study visit 1)
  Measured at baseline and 30 min post intervention to assess change in response. (0=no pain, 100=most pain)
  * Heat Pain - 1) A slowly increasing heat stimulus (44°C, 46°C, and 48°C) will be delivered; 2) a series of 5 heat pulses (about 2 sec) will be given and pain will be rated (0-100)
  * Touch Test Pain. Von Frey filament will be tapped on knee and hand and asked to rate the pain (0-100) after a single tap, and after 10 consecutive taps
  * Pressure Pain Threshold. A slowly increasing pressure will be applied on forearm and shoulder with a probe (Algomed) till pain is felt. Then constant pressure will be applied till the sensation first becomes painful to assess threshold in kilopascals
  * Combined Pressure and Cold Pain. Hand will be immersed in cold water (10°C). After 30 sec, pain intensity will be rated (0-100). Hand will be kept in cold water for another 30 sec and then the pressure pain test will be performed, and first instance of pain due to pressure will be assessed
Quantitative sensory testing (QST) | Study visit 2 will occur at least 5-7 days after the first visit
  Measured at baseline and 30 min post intervention to assess change in response. (0=no pain, 100=most pain)
  * Heat Pain - 1) A slowly increasing heat stimulus (44°C, 46°C, and 48°C) will be delivered; 2) a series of 5 heat pulses (about 2 sec) will be given and pain will be rated (0-100)
  * Touch Test Pain. Von Frey filament will be tapped on knee and hand and asked to rate the pain (0-100) after a single tap, and after 10 consecutive taps
  * Pressure Pain Threshold. A slowly increasing pressure will be applied on forearm and shoulder with a probe (Algomed) till pain is felt. Then constant pressure will be applied till the sensation first becomes painful to assess threshold in kilopascals
  * Combined Pressure and Cold Pain. Hand will be immersed in cold water (10°C). After 30 sec, pain intensity will be rated (0-100). Hand will be kept in cold water for another 30 sec and then the pressure pain test will be performed, and first instance of pain due to pressure will be assessed

SECONDARY OUTCOMES:
McGill Pain Questionnaire-Short Form | At baseline (study visit 1)
  15 descriptors (11 sensory; 4 affective) using an intensity scaled ranging from 0-3 on pain scale (0 = no pain, 1 = mild pain, 2 = moderate pain or 3 = severe pain)
McGill Pain Questionnaire-Short Form | Study visit 2 will occur at least 5-7 days after the first visit
  15 descriptors (11 sensory; 4 affective) using an intensity scaled ranging from 0-3 on pain scale (0 = no pain, 1 = mild pain, 2 = moderate pain or 3 = severe pain)
Measuring endogenous opioid peptides in plasma and peripheral leukocytes | At baseline (study visit 1)
  20 ml blood will be drawn to isolate plasma and peripheral leukocytes

CONTACTS AND LOCATIONS:
Overall Officials: Saurabh Aggarwal, MD., PhD, Principal Investigator — Florida International University
Locations (1):
- Ambulatory Care Center, Florida International University, Miami, Florida, United States